CLINICAL TRIAL: NCT03260374
Title: Objective Measures in Cochlear Implant in Children and Its Correlation to Outcome
Brief Title: Objective Measures in Cochlear Implant
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dina Mohamed, director, Assiut University
Other Study IDs: OMCI
Record Dates: First submitted 2017-08-20; First posted 2017-08-24 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Sensorineural Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- children with cochlear implant: 30 subjects whose age ranges from 2-6 years old who are implanted with Medel multichannel cochlear implant male and female will be included and will undergo:-
  * Electric compound action potential
  * Electric stapedial reflex threshold
  * Electric auditory brain stem response
  Interventions: Device: Electric compound action potential; Device: electric stapedial reflex threshold; Device: electric auditory brain stem response

INTERVENTIONS:
Device: Electric compound action potential — The electrically evoked compound action potentials, which are closely related to the electrically evoked brainstem responses, would also show a similar correlation with the behavioral threshold. Determining threshold levels requires subjective responses to a series of sophisticated psychophysical percepts. This is often difficult for cochlear implant patients. However, the neural response telemetry system renders possible the measurement of the compound action potential threshold .
Device: electric stapedial reflex threshold — electric stapedial reflex threshold measurements are performed using the same software platform and electrical stimulus utilized for fitting the cochlear implant . Thus, stimulus parameters, including pulse duration and repetition rate, can be identical to those used to obtain behavioral judgments for psychophysical levels
Device: electric auditory brain stem response — For most implant recipients , even the first introduction of electric stimulation from a cochlear implant evokes activity in the auditory brainstem , which can be measured as clear electric auditory brain stem response waveforms . Therefore the electric auditory brain stem response test can be used in the functional evaluation of the auditory system between the time of initial implant activation and after chronic cochlear implant use

SUMMARY:
One of the main factors affecting the ability to maximize the full potential of a cochlear implant is an accurate map.The goal of mapping is to enable cochlear implant recipients to perceive a desired range of acoustic signals. The process includes programming of the minimum and the maximum stimulation levels that are based on subjective measurements of thresholds and the most comfortable level . The use of objective measures in the CI process has greatly contributed to the definition of the dynamic field, as they provide specific values that serve as the basis for the start of the mapping process, especially in cases of infants and young children. Some examples of these measures are electrically evoked stapedius reflex threshold , neural response telemetry , brainstem auditory evoked potential , and P300, among others.

DETAILED DESCRIPTION:
In adult Cochlear implant users, programming is a relatively straightforward task as psychophysical measurements can be explained, and patients quickly understand the link between the mapping process and the output of their system . In young children or infants, the mapping process is more complex, especially comfort levels. Setting the threshold level requires the child to respond to the presence or the absence of a sound. Although the same techniques are used in setting the comfort level, the child is now required to make a judgment about the sound beyond its simple presence or absence. Young children often lack the attention span, patience, and cognitive and language skills necessary to perform these tasks with good reliability and repeatability .The use of objective measures in the CI process has greatly contributed to the definition of the dynamic field, as they provide specific values that serve as the basis for the start of the mapping process, especially in cases of infants and young children. Some examples of these measures are electrically evoked stapedius reflex threshold , neural response telemetry , brainstem auditory evoked potential , and P300, among others.The electrically evoked compound action potentials, which are closely related to the electrically evoked brainstem responses, would also show a similar correlation with the behavioral threshold . Determining threshold levels requires subjective responses to a series of sophisticated psychophysical percepts. This is often difficult for cochlear implant patients. However, the neural response telemetry system renders possible the measurement of the compound action potential threshold . Electric stapedial reflex threshold measurements are performed using the same software platform and electrical stimulus utilized for fitting the cochlear implant . Thus, stimulus parameters, including pulse duration and repetition rate, can be identical to those used to obtain behavioral judgments for psychophysical levels .For most implant recipients , even the first introduction of electric stimulation from a cochlear implant evokes activity in the auditory brainstem , which can be measured as clear electric auditory brain stem response waveforms . Therefore this test can be used in the functional evaluation of the auditory system between the time of initial implant activation and after chronic cochlear implant use.

ELIGIBILITY:
Inclusion Criteria:

* children implanted with Medel multichannel cochlear implant

Exclusion Criteria:

* • Any middle ear problem

  * Any technical problems with the cochlear implant device

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children with sensorineural hearing loss implanted with Medel multi-channel cochlear implant aged 2-6 years
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2019-08-31 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Arabic language test | 2 years
  Speech and language assessment in children with cochlear implant